CLINICAL TRIAL: NCT05046977
Title: Double Osteotomy for Deformity Correction In Pyle Disease: Comparative Study
Brief Title: Double Osteotomy for Deformity Correction in Pyle Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Sherwan Ahmed Ali Hamawandi, Assistant professor of orthopedic surgery, Hawler Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMU/Sherwan14
Record Dates: First submitted 2021-09-12; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Pyle Disease
Keywords: Pyle disease; Genu valgus; Double Osteotomy; Deformity analysis; Functional outcome
MeSH Terms: conditions — Pyle disease; Genu Valgum | interventions — Osteotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single tibial osteotomy (Active Comparator): Single tibial osteotomy done to achieve correction
  Interventions: Procedure: Single osteotomy
- Double tibial osteotomy (Active Comparator): Double tibial osteotomy done to achieve correction
  Interventions: Procedure: Double Osteotomy

INTERVENTIONS:
Procedure: Single osteotomy — Single tibial osteotomy
  Arms: Single tibial osteotomy
Procedure: Double Osteotomy — Double Tibial Osteotomy
  Arms: Double tibial osteotomy

SUMMARY:
Leg deformity is one of the features of Pyle disease( metaphyseal dysplasia). Correction of valgus deformity of the leg can be done after deformity analysis by double osteotomy so this study showed how double osteotomy can lead to better results than single osteotomy.

ELIGIBILITY:
Inclusion Criteria:

* Pyle Disease

Exclusion Criteria:

1. Smoking
2. Diabets Mellitus
3. Previous surgery on the limbs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2021-09-20 (Estimated); Primary Completion 2022-09-20 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Mechanical axis of lower limbs | This mechanical axes were assessed one year after surgery
  This will determine how much the mechanical axes of the lower limbs were diverted from the normal values. We asked for lower limb radiograph in both Anteroposterior and lateral views and we measure the mechanical axes of the whole lower limb and that of tibial and measures how much the proximal medial tibial angle and compared with normal values
Knee injury and Osteoarthritis outcome score | This score was assessed one year post-operatively
  This score involves six sections from zero score to 100. The more score is better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Hawler medical University, Erbil, Iraq